CLINICAL TRIAL: NCT02436850
Title: Bed Side Thoracentesis Among Non-Ventilated Patients With Respiratory Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ori Galante, Dr. Ori Galante, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0116-15-CTIL
Record Dates: First submitted 2015-04-20; First posted 2015-05-07 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Instability
Keywords: Thoracentesis; Pocket Ultrasound Device; Ultrasound; Soroka University Medical Center; Physical Examination; Ethical Committee
MeSH Terms: interventions — Thoracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive large volume thoracentesis.
  Interventions: Procedure: Thoracentesis
- Control group (No Intervention): The control group will be taped with an 18 gauge and 20 gauge venflons and drain will not be placed.

INTERVENTIONS:
Procedure: Thoracentesis — An invasive procedure to remove fluid or air from the pleural space for diagnostic or therapeutic purposes.
  Arms: Intervention group

SUMMARY:
The purpose of the trial is to evaluate the effectiveness of moderate to large volume thoracentesis (TC) in non-ventilated patients in Internal Medicine admitted due to, or suffer from respiratory instability. This is a prospective, double-center, randomized clinical trial. This is a stage 1 pilot trial aimed to provide better understanding on the study population and study groups. This trial will comprise a total of 60 patients, 30 subjects on the intervention group and an equal number on the control group. The results of this pilot trial will be to design a larger trial and calculate a required sample size.

DETAILED DESCRIPTION:
The prevalence of pleural effusion is high among medical patients, reaching 62% among Medical ICU patients. Often clinicians are standing in front of a symptomatic respiratory patient with moderate or large pleural effusion. The clinical question whether TC will be beneficial for the patient with respiratory compromise is yet to be shown. There are few, small scale studies on the benefit of pleural effusion thoracentesis. Only one study found sustained effect of thoracentesis on oxygenation among 10 patients on mechanical ventilation. Lung function was found to improve after TC among patients with paradoxical movement of hemidiaphragm, and relief of dyspnea after large pleural effusion TC was demonstrated as well. No study to date, as the investigators know, on the benefit of TC, was done on non-ventilated, ward patients with moderate to large pleural effusion. Also, no studies to date showed any improved clinical outcome of this procedure.

Although ultrasound guided TC is a safer mode than blinded TC, complications as pneumothorax, pain, shortness of breath, cough, bleeding, hematoma, and re-expansion pulmonary edema may result from TC. Although no consensus exist regarding the benefit of TC still this procedure is common among ventilated and non-ventilated patients. The investigators seek to find whether there is clinical benefit for TC, among non-ventilated, ward patients with moderate to large pleural effusion. For this purpose the investigators aim to conduct a prospective randomized trial.

In this study the investigators aim to compare outcomes as: hospital length of stay, vital signs and wellbeing, utilization of imaging modalities and readmission rates among patients who had therapeutic TC compared to those who had not. Also the investigators would like to try and predict the amount of pleural effusion from the ultrasound imaging as well as to find the added value of point of care US screening of pleural effusion on top of routine Xr among patients with respiratory instability.

To the best of the investigators' knowledge, no prospective randomized study to date has compared the strategy of TC to none among non-ventilated ward patients with respiratory complains.

This is a prospective, double-center, randomized clinical trial. This is a stage 1 pilot trial aimed to provide better understanding on the study population and study groups. This trial will comprise a total of 60 patients, 30 subjects on the intervention group and an equal number on the control group. The results of this pilot trial will be to design a larger trial and calculate a required sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to internal ward
2. Patients with moderate to large pleural effusion per ultrasound as defined under Eligibility section below
3. At least of the following findings:

   * Dyspnea on admission notes
   * Tachypnea (RR >18 pm)
   * Desaturation (saturation<88%)
   * Admission diagnosis of CHF exacerbation or any uncontrolled heart failure,
   * Effort dyspnea per history,
   * Acute or subacute (last two weeks) need for oxygen supplement or Noninvasive ventilation.
   * Admission diagnosis of pulmonary edema or pulmonary congestion
   * Hypoxemia (PaO2<60mmHg)
   * Pleuritic chest pain

Exclusion Criteria:

1. Subject currently enrolled in another investigational study
2. Patients on mechanical ventilation
3. Patients with coagulopathy (known or with any prolongation of PTT, PT, fibrinogen<200, platelets <100000)
4. Patients with cognitive impairment who cannot sign informed consent
5. Patients with sepsis or fever and pneumonia and suspected empyema
6. Patients with any previous surgeries to the lungs
7. Patients whom the primary team call for therapeutic TC.
8. Patients with less than moderate amount of pleural effusion (see Eligibility criteria)
9. Palliative patients
10. Pregnant patients
11. On any current anticoagulation therapy or with any abnormal coagulation study.
12. Patients with septations or cavitation in pleural space (visible on US

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | 12 months

SECONDARY OUTCOMES:
Vital signs and wellbeing questionnaire | 12 months
Readmission rates | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Fartoukh M, Azoulay E, Galliot R, Le Gall JR, Baud F, Chevret S, Schlemmer B. Clinically documented pleural effusions in medical ICU patients: how useful is routine thoracentesis? Chest. 2002 Jan;121(1):178-84. doi: 10.1378/chest.121.1.178. PMID 11796448
- [Background] Mattison LE, Coppage L, Alderman DF, Herlong JO, Sahn SA. Pleural effusions in the medical ICU: prevalence, causes, and clinical implications. Chest. 1997 Apr;111(4):1018-23. doi: 10.1378/chest.111.4.1018. PMID 9106583
- [Background] Walden AP, Garrard CS, Salmon J. Sustained effects of thoracocentesis on oxygenation in mechanically ventilated patients. Respirology. 2010 Aug;15(6):986-92. doi: 10.1111/j.1440-1843.2010.01810.x. Epub 2010 Jul 20. PMID 20646244
- [Background] Collins TR, Sahn SA. Thoracocentesis. Clinical value, complications, technical problems, and patient experience. Chest. 1987 Jun;91(6):817-22. doi: 10.1378/chest.91.6.817. PMID 3581930
- [Background] Wang LM, Cherng JM, Wang JS. Improved lung function after thoracocentesis in patients with paradoxical movement of a hemidiaphragm secondary to a large pleural effusion. Respirology. 2007 Sep;12(5):719-23. doi: 10.1111/j.1440-1843.2007.01124.x. PMID 17875061
- [Background] Estenne M, Yernault JC, De Troyer A. Mechanism of relief of dyspnea after thoracocentesis in patients with large pleural effusions. Am J Med. 1983 May;74(5):813-9. doi: 10.1016/0002-9343(83)91072-0. PMID 6837605
- [Background] Jones PW, Moyers JP, Rogers JT, Rodriguez RM, Lee YC, Light RW. Ultrasound-guided thoracentesis: is it a safer method? Chest. 2003 Feb;123(2):418-23. doi: 10.1378/chest.123.2.418. PMID 12576360
- [Background] Perazzo A, Gatto P, Barlascini C, Ferrari-Bravo M, Nicolini A. Can ultrasound guidance reduce the risk of pneumothorax following thoracentesis? J Bras Pneumol. 2014 Jan-Feb;40(1):6-12. doi: 10.1590/S1806-37132014000100002. PMID 24626264
- [Background] Eibenberger KL, Dock WI, Ammann ME, Dorffner R, Hormann MF, Grabenwoger F. Quantification of pleural effusions: sonography versus radiography. Radiology. 1994 Jun;191(3):681-4. doi: 10.1148/radiology.191.3.8184046.
- [Background] Lichtenstein D, Hulot JS, Rabiller A, Tostivint I, Meziere G. Feasibility and safety of ultrasound-aided thoracentesis in mechanically ventilated patients. Intensive Care Med. 1999 Sep;25(9):955-8. doi: 10.1007/s001340050988. PMID 10501751
- [Background] Balik M, Plasil P, Waldauf P, Pazout J, Fric M, Otahal M, Pachl J. Ultrasound estimation of volume of pleural fluid in mechanically ventilated patients. Intensive Care Med. 2006 Feb;32(2):318. doi: 10.1007/s00134-005-0024-2. Epub 2006 Jan 24. PMID 16432674
- [Background] Vignon P, Chastagner C, Berkane V, Chardac E, Francois B, Normand S, Bonnivard M, Clavel M, Pichon N, Preux PM, Maubon A, Gastinne H. Quantitative assessment of pleural effusion in critically ill patients by means of ultrasonography. Crit Care Med. 2005 Aug;33(8):1757-63. doi: 10.1097/01.ccm.0000171532.02639.08. PMID 16096453
- [Background] Roch A, Bojan M, Michelet P, Romain F, Bregeon F, Papazian L, Auffray JP. Usefulness of ultrasonography in predicting pleural effusions > 500 mL in patients receiving mechanical ventilation. Chest. 2005 Jan;127(1):224-32. doi: 10.1378/chest.127.1.224. PMID 15653988
- [Background] Feller-Kopman D, Walkey A, Berkowitz D, Ernst A. The relationship of pleural pressure to symptom development during therapeutic thoracentesis. Chest. 2006 Jun;129(6):1556-60. doi: 10.1378/chest.129.6.1556. PMID 16778274